CLINICAL TRIAL: NCT06003660
Title: BrainFlavor: Brain Neuronal Networks and Chemosensory and Trigeminal Functions in Allogeneic Hematopoietic Stem Cell Transplantation - a Prospective Cohort-study
Brief Title: Brain Neuronal Networks, Chemosensory and Trigeminal Functions in Allo-HSCT
Status: Recruiting | Type: Observational
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Per Ole Iversen, MD, Professor, University of Oslo
Other Study IDs: 282886
Record Dates: First submitted 2023-08-10; First posted 2023-08-22 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Adult recipients of allo-HCST.
- Controls: Healthy adult subjects

SUMMARY:
The goal of this prospective, cohort study is to learn about smell, taste and trigeminal dysfunction in patients receiving allogeneic hematopoietic stem cell transplantation (allo-HSCT). The research team hypothesizes that treatment with allo-HSCT will induce:

* Distortion of taste and smell and trigeminal functions like cooling, tingling, and burning sensations.
* Reduced saliva production leading to oral dryness and dental caries.
* Changes in the connectivity of the taste-, smell- and pain-cortical brain regions.

DETAILED DESCRIPTION:
Participants will undergo various tests:

* Smell function assessment with Sniffin' Sticks.
* Taste function assessment with Taste Strips.
* Oral trigeminal function assessment with von Frey filaments .
* Salivary assessment with the Summated Xerostomia Inventory-Dutch questionnaire.
* Salivary flow will be measured using salivary flow rate - stimulated whole saliva (SWS).
* A clinical oral examination will be done to obtain a Clinical Oral Dryness Score.
* Qualitative smell, taste and trigeminal dysfunction will be assessed using a questionnaire.
* Radiological and clinical examinations will be performed to evaluate dental and oral mucosal status.
* Quality of life using questionnaire.
* Nutritional status using questionnaire.
* Magnetic resonance imaging of the brain will be taken to capture regions-of-interest for the three different networks of interest; (i) the gustatory network reflecting changes in taste perception, (ii) the olfactory network, related to the changes in smell, and (iii) the pain matrix reflecting pain.

There will be a comparisons between the patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

• patients receiving myeloablative conditioning for a first-time allo-HSCT and diagnosed with either a leukemia or a myelodysplastic syndrome

Exclusion Criteria:

* disorders affecting the oral cavity including poor tooth-status
* those using drugs affecting the gustatory/olfactory functions
* those with brain disorders
* those who have a chronic disorder affecting the immune system, have cancer or who are pregnant.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients receiving myeloablative conditioning for a first-time allo-HSCT and diagnosed with either a leukemia or a myelodysplastic syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Olfactory (smell) function | 1 year
  Odour pens of the Sniffin' Sticks (Burghart Messtechnik, Wedel, Germany) will be used to test olfactory function (TDI). Scores will range from 0 - 48 where score ≤ 16.5 = anosmia (no sense of smell), score 16.6 - 30.5 = hyposmia (reduced sense of smell) and score >30.5 = normosmia (normal sense of smell)
Self-reported olfactory (smell) function | 1 year
  Self-reported smell function will be assessed using a visual analogue scale (VAS) ranging from 0-10 where 0 indicates no smell function and 10 very good smell function.
Gustatory (taste) function | 1 year
  Taste function will be evaluated by using taste strips ("Taste Strips "Burghart Messtechnik, Wedel, Germany) with four basic taste qualities (sweet, sour, salty and bitter) in 4 different concentrations each. Scores will range from 0 - 16 where 0 = ageusia (no sense of taste), 1 - 9 = hypogeusia (reduced sense of smell) and 10 - 16 = normogeusia (normal sense of taste)
Self-reported gustatory (taste) function | 1 year
  Self-reported taste function will be assessed using a visual analogue scale (VAS) ranging from 0-10 where 0 indicates no taste function and 10 very good taste function.
Oral pain assessment | 1 year
  Oral pain perception will be assessed by von Frey filaments. Scores will range from 0 -10 on a visual analogue scale (VAS) where 0 indicates no pain and 10 severe pain.
Self-reported oral pain assessment | 1 year
  Self-reported oral pain will be assessed using a visual analogue scale (VAS) ranging from 0-10 where 0 indicates no oral pain and 10 severe oral pain.
Functional brain connectivity | 1 year
  Functional connectivity analysis (fMRI) of three different networks of interest: (i) the olfactory network (ii) the gustatory, and (iii) the pain matrix. There are no specified quantitative units for these measurements.

SECONDARY OUTCOMES:
Measured oral dryness | 1 year
  Saliva production will be measured using salivary flow rate - stimulated whole saliva (SWS). Hyposalivation is defined as a salivary secretion rate of ≤0.7 mL/min for SWS.
Clinical oral dryness | 1 year
  Clinical oral dryness will be assessed using Clinical Oral Dryness Score (CODS). Scores will range from 0 to 10 points. Score 1-3 is considered mild oral dryness, 4-6 moderate and 7-10 severe oral dryness.
Self-reported oral dryness | 1 year
  Self-reported oral dryness will be assessed using the Xerostomia Inventory (XI) questionnaire. Scores will range from 11 to 55 points, with values <14 considered as normal.
Oral mucosal status | 1 year
  Oral mucosal status will be evaluated using mucosal-plaque index (MPS). Scores will range from 2 - 8 where 2 - 4 = good/acceptable, 5 - 6 = no acceptable and 7 - 8 = poor status
Oral mucositis status | 1 year
  Oral mucosal status will be evaluated using the WHO mucositis grading ranging form 0 - 4 where 0 = no oral mucositis, 1 = erythema and soreness, 2 = ulcers, able to eat solids, 3 = ulcers, requires a liquid diet (due to mucositis), 4 = ulcers, alimentation not possible (due to mucositis)
Nutritional status | 1 year
  Nutritional status will be evaluated using the Nutrition Risk Screening 2002 form. Scores range from 0-6. Patients with a score < 3 is considered to be of no nutritional risk. Patients with a score ≥ 3 is considered to be in nutritional risk.
Quality of life evaluation | 1 year
  Quality of life will be assessed using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). Scores range from 0-100. A high score indicates better quality of life and a low score indicates a worse quality of life.
Oral health-related quality of life evaluation | 1 year
  Oral health-related quality of life will be assessed using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. Scores range from 0-56. A high score indicates worse oral health-related quality of life, while a low score indicates better.

CONTACTS AND LOCATIONS:
Overall Officials: Per Ole Iversen, phd, Study Director — University of Oslo
Locations (1):
- University of Oslo, Oslo, Oslo County, Norway